CLINICAL TRIAL: NCT02809521
Title: Increasing Spontaneous Non-exercise Activity (The Sitting Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GFHNRC149
Record Dates: First submitted 2016-06-17; First posted 2016-06-22 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Activity Liking (Other): Subjects will look at images of people doing different types of activities (e.g., walking, skiing, watching television) and rate their liking of the activity.
  Interventions: Other: Activity Liking

INTERVENTIONS:
Other: Activity Liking

SUMMARY:
The purpose of the study is to see if one's liking and awareness of different types of activities is related to one's activity pattern.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary lifestyle

Exclusion Criteria:

* 5% weight loss within the past 2 months
* Active job or lifestyle
* Participation in an exercise program
* Pregnant and/or lactating
* Uncontrolled hypertension
* Alcohol or drug abuse
* Presence of acute illness
* Major limitation of physical movement

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in liking of activity | Baseline, week 1, week 2
  Visual Analog Scale rating and operant responses for sedentary and physical activities

CONTACTS AND LOCATIONS:
Overall Officials: Shanon Casperson, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No